CLINICAL TRIAL: NCT03114215
Title: Effect of MD1003 in Amyotrophic Lateral Sclerosis: a Randomized Double Blind Placebo Controlled Pilot Study
Brief Title: Effect of MD1003 in Amyotrophic Lateral Sclerosis
Acronym: MD1003-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MD1003CT2015-02-ALS
Record Dates: First submitted 2017-03-28; First posted 2017-04-14 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: Biotin; MD1003; ALSFRS-R
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Biotin

STUDY DESIGN:
Intervention Model Description: The primary objective of the study is to evaluate the safety of biotin at 300 mg/day over placebo in patients with amyotrophic lateral sclerosis.
  This is a 6-month double blind randomized 2:1 placebo-controlled study with two arms (placebo, biotin 300 mg/day). The study will be followed by a 6-month extension phase during which all patients will receive biotin 300 mg/day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MD1003 (Active Comparator): The investigational drug will consist in capsules of 100 mg biotin and excipients (lactose, magnesium stearate, croscarmellose sodium, Silica) tid during 12 months
  Interventions: Drug: MD1003
- PLACEBO (Placebo Comparator): This formulation consists in lactose powder and other excipients (magnesium stearate, croscarmellose sodium, Silica) as placebo, tid during 6 months and then switch to MD1003 tid during 6 additional months.
  Interventions: Drug: MD1003; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: MD1003 — capsules 100mg 3 times per day
  Other Names: BIOTIN
Drug: Placebo oral capsule — capsules 100mg lactose 3 times per day
  Arms: PLACEBO

SUMMARY:
This is a 6-month double blind randomized 2:1 placebo-controlled study with two arms (placebo, biotin 300 mg/day). The study will be followed by a 6-month extension phase during which all patients will receive biotin 300 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25 to 80 years, inclusive
* Male or female subjects with probable or confirmed ALS (revised international El Escorial criteria, Forbes et al., 2001).
* Patients presenting first motor deficits due to ALS for a maximum of three years at the first consultation in an ALS centre.
* Patients monitored for at least 6 months in an ALS centre or for whom the previous monitoring parameters are available (excepted for MIP and SNIP).
* Patients who have lost at least 5 points on the ALSFRS-R (ALS functional rating scale) during the last 12 months or at least 2 points during the preceding 6 months
* Patients who have been treated with riluzole for at least 3 months at a stable dose. In case of intolerance to this product or refusal for this treatment, patients who have not been treated with riluzole for at least 1 month before inclusion
* For patients with spinal form (onset of the disease affecting limbs) or respiratory form, slow vital capacity > 60% of predicted value.
* For patients with a bulbar form, slow vital capacity > 60% of theoretical value or, if spirometry not assessable (severe bulbar disability), patient should not have significant abnormality in both nocturnal capnography and nocturnal oximetry (median pCO2 (carbon dioxide partial pressure ) < 52 mmHg, SaO2 (arterial oxygen saturation ) < 90% less than 5% of the time during night) less than 3 months prior inclusion.
* Patients who are willing to give written consent (or oral consent in the presence of a trusted person if the patient is no longer able to write)
* Patients likely to be able to participate in all scheduled evaluation and complete all required study procedures (except for spirometry in bulbar patients with severe disability).

Exclusion Criteria:

* Patients on non-invasive ventilation for respiratory insufficiency due to ALS for more than 10 hours a day
* Patients with an ALSFRS-R score at inclusion of < 20 (maximum score without disability = 48)
* Patients who have lost less than 5 points on the ALSFRS-R during the last year or less than 2 points during the preceding 6 months
* Patients with a gastrostomy
* Patients who have lost more than 15% of their reference weight (defined as weight before disease onset)
* Patient with dyspnoea at rest or with the least effort (score < 3 on the dyspnoea item of the ALSFRS-R)
* Patients with dementia
* Patient with severe or rapidly progressive form of ALS for whom the investigator estimates the life expectancy less than 3 months
* Patients with another progressive disease that has not been stabilized at the time of inclusion
* Patients with cancer, except basal cell carcinoma, for less than 5 years, or who require continuous treatment for cancer even if it is older
* Pregnant women.
* Subject who are not covered by a social security scheme.
* Subject under temporary or permanent Judicial Protection.
* Contraception: Both male subjects, and female subjects who are not either surgically sterile (tubal ligation/obstruction or removal of ovaries or uterus) or post-menopausal (no spontaneous menstrual periods for at least one year confirmed by a negative hormone panel), must commit to using two highly effective method of birth control for the duration of the study and for two months after the treatment termination.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recording of adverse events | 6 months
  All adverse events in two groups will be recorded.
Laboratory testing (haematology and biochemistry panel) | 6 months
  * RBC (red blood cell), WBC (white blood cell ), platelets
  * Ferritin, CPK (creatine phosphokinase )
  * Electrolytes, creatinine, glycaemia
  * AST (aspartate aminotransferase ), ALT (alanine aminotransferase) , bilirubin, GGT (gamma-glutamyltransferase), alkaline phosphatase
  * Triglyceride, cholesterol
  * Haemostasis: APPT (activated partial thromboplastin time), PT (prothrombin time )

SECONDARY OUTCOMES:
Motor disability | 6 months
  this is evaluated using the ALSFRS-R scale (score of 48 points). Among the criteria used to evaluate the severity of ALS, the rate of the decline in the ALSFRS-R is the one that correlates most closely with the risk of death (Kimura et al., 2006).
Severity | 6 months
  The severity of the disease defined as the ratio between the number of points lost on the ALSFRS-R score and the number of months that have elapsed (Kollewe et al., 2008).
Slow vital capacity (SVC) | 6 months
  in liters
Maximal inspiratory pressure (MIP) | 6 months
  in cm H2O
Sniff nasal inspiratory pressure (SNIP) | 6 months
  in cm H20
Weight | 6 months
  weight in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Gui De Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juntas-Morales R, Pageot N, Bendarraz A, Alphandery S, Sedel F, Seigle S, Camu W. High-dose pharmaceutical grade biotin (MD1003) in amyotrophic lateral sclerosis: A pilot study. EClinicalMedicine. 2020 Jan 27;19:100254. doi: 10.1016/j.eclinm.2019.100254. eCollection 2020 Feb. PMID 32140672